CLINICAL TRIAL: NCT07052617
Title: A Multicentric Observational Study Examining How Different CRRT Modalities, Dosing Strategies, and Timing Impact Kidney Recovery and the Development of Prolonged Kidney Dysfunction (Acute Kidney Disease) in Critically Ill Patients
Brief Title: Impact of Different CRRT Modalities, Dosing Strategies, and Timing on Kidney Recovery and Prolonged Kidney Dysfunction
Acronym: KARMA
Status: Not yet recruiting | Type: Observational
Sponsor: Croatian Society for Organ Support (Other)
Responsible Party: Principal Investigator, Vedran Premuzic, Assistant Professor, M.D., Ph.D., Croatian Society for Organ Support
Other Study IDs: 02/013AG; CSOS2025 (Other: Croatian Society for Organ Support)
Record Dates: First submitted 2025-06-21; First posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Acute Kidney Disease; Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Continuos renal replacement therapy — Different modalities of CRRT: continuous veno-venous hemofiltration; continuous veno-venous hemodialysis and continuous veno-venous hemodiafiltration Different doses of CRRT: low effluent dose (<15 ml/kg/h); medium-low effluent dose (15-25 ml/kg/h); standard effluent dose (25-30 ml/kg/h); high effluent dose (>30 ml/kg/h

SUMMARY:
KARMA study is a hospital-based research study looking at how different ways of delivering kidney support therapy (CRRT) affect patients who are critically ill. In some cases, the kidneys may temporarily stop working in very sick patients, and machines are used to filter the blood. This study is exploring whether the way the investigators use these machines - how early to start, how much treatment to give, and what type to choose - makes a difference in how well the kidneys recover. By learning from many hospitals and hundreds of patients, KARMA hopes to improve treatment choices and help patients regain their kidney function faster.

ELIGIBILITY:
Inclusion Criteria:

* Acute kidney injury
* ICU administration

Exclusion Criteria:

* Pre-existing CKD (GFR < 30 ml/min/1,73m2)
* Chronic dialysis-dependent end-stage renal failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: By analyzing the variation in therapeutic approaches across centers-including convection- and diffusion-based techniques, dose intensity, and initiation thresholds-KARMA study aims to identify best practices that promote renal recovery and reduce the transition to acute kidney disease. The study integrates clinical, biochemical, and outcome metrics to support a precision medicine framework in critical care nephrology and in critically ill patients with acute kidney injury.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2025-09-25 (Estimated); Primary Completion 2026-09-25 (Estimated); Study Completion 2026-12-25 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with AKD | 90 days
  Percentage of patients with AKD divided by subgroups regarding AKI etiology

SECONDARY OUTCOMES:
Durations and severity of AKD, free days of CRRT and kidney recovery | 90 days
  AKD duration in days AKD severity described and compared by AKI stages Patients with AKD divided by subgroups regarding indication for CRRT (fluid overload, electrolyte disturbances, metabolic acidosis, uremia, oliguria/anuria) and CRRT dose (ml/kg/hour) CRRT free days during ICU Kidney recovery/stage of CKD/dialysis dependency

IPD SHARING:
Plan to Share IPD: Yes
Specific IPD including information like a participant's age, sex, treatment received, and specific outcomes will be shared
Supporting Information: Study Protocol
Time Frame: Start date: December 25, 2025 End date: October 25, 2026